CLINICAL TRIAL: NCT03950960
Title: An Open-label, Single-Sequence, 2-Treatment Period Study to Investigate the Effects of Cytochrome P450 3A4 Inhibition by Itraconazole on the Pharmacokinetics of BMS-986256 in Healthy Participants
Brief Title: A Study to Investigate the Effects of Itraconazole on the Pharmacokinetics of BMS-986256 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM026-020
Record Dates: First submitted 2019-05-14; First posted 2019-05-15 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Healthy Participants
Keywords: Cytochrome P450 3A4 Inhibition
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986256 +Itraconazole (Experimental)
  Interventions: Drug: BMS-986256; Drug: Itraconazole

INTERVENTIONS:
Drug: BMS-986256 — Specified dose on specified days
Drug: Itraconazole — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the effect of cytochrome P450 3A4 inhibition by Itraconazole on the pharmacokinetics of BMS-986256.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy participant, defined as having no clinically significant active or ongoing medical condition, physical examination abnormality, abnormal ECG finding, and abnormal clinical laboratory determinations that in the opinion of the Investigator would compromise the conduct, results, or interpretation of the study findings
* A negative QuantiFERON®-TB Gold test result at screening or documentation of a negative result within 3 months of the screening visit
* Weight greater than or equal to (>=) 50 kilogram (kg) and body mass index between 18.0 and 32.0 kilogram per meter square (kg/m^2) inclusive at screening

Exclusion Criteria:

* Prior exposure to BMS-986256
* Previous investigational drug or placebo exposure within 6 weeks before nonbiologic study drug administration or 12 weeks before biologic study drug administration
* History or presence of malignancy including hematological malignancies. However, participants with a history of basal cell or squamous cell carcinoma that has been completely and successfully treated with no evidence of recurrence may not be excluded, at the discretion of the investigator

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of BMS-986256 | After single dose on Days 1 and 29
Area Under the Plasma Concentration-time Curve from Time Zero to Time of Last Quantifiable Concentration (AUC[0-T]) of BMS986256 | After single dose on Days 1 and 29
Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC[INF]) of BMS-986256 | After single dose on Days 1 and 29

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | From the time of study treatment administration through the final study visit (Up to 55 days)
Percentage of Participants with Serious Adverse Events (SAEs) | From the time ICF is signed through 30 days post dose, or the final study visit (Up to 60 days)
Percentage of Participants with Vital Signs, Electrocardiograms (ECGs), and Physical Examinations Abnormalities | From screening to follow-up (Up to 55 days)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences - Lenexa, Lenexa, Kansas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm